CLINICAL TRIAL: NCT06511050
Title: Investigating the Effects of Lumbrokinase in Adults With Long Covid, Post-treatment Lyme Disease Syndrome, and Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Brief Title: Lumbrokinase for Adults With Long Covid, Post-treatment Lyme Disease Syndrome, and Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Columbia University (Other); PolyBio Research Foundation (Other)
Responsible Party: Principal Investigator, David Putrino, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-24-00154
Record Dates: First submitted 2024-07-16; First posted 2024-07-19 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-09

CONDITIONS: Long Covid; Post-treatment Lyme Disease Syndrome; Chronic Fatigue Syndrome; Myalgic Encephalomyelitis
Keywords: Long Covid; Lyme Disease; ME/CFS; Lumbrokinase; Post-treatment Lyme disease syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Post-Lyme Disease Syndrome; Fatigue Syndrome, Chronic; Lyme Disease | interventions — lumbrokinase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Long Covid (Experimental): Boluoke® brand lumbrokinase capsules, 300,000 functional units (FUs) twice per day, daily for 6 weeks.
  Interventions: Dietary Supplement: Lumbrokinase
- Post-treatment Lyme Disease Syndrome (Experimental): Boluoke® brand lumbrokinase capsules, 300,000 functional units (FUs) twice per day, daily for 6 weeks.
  Interventions: Dietary Supplement: Lumbrokinase
- Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (Experimental): Boluoke® brand lumbrokinase capsules, 300,000 functional units (FUs) twice per day, daily for 6 weeks.
  Interventions: Dietary Supplement: Lumbrokinase

INTERVENTIONS:
Dietary Supplement: Lumbrokinase — Boluoke® brand lumbrokinase capsules will be taken daily for 6 weeks.
  Other Names: Boluoke® Lumbrokinase

SUMMARY:
This will be a pilot multi-arm clinical trial investigating the feasibility of Lumbrokinase (LK) as an intervention in three clinical cohorts:

* Long Covid (LC)
* Post-treatment Lyme disease syndrome (PTLDS)
* Myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS)

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* Aged 18+
* Baseline EQ-VAS ≤70; EQ-VAS before the index infection ≥80 (this information is collected as part of the baseline survey).
* Diagnosed with only one of the following conditions:
* Long Covid
* Documented clinical history of confirmed or suspected acute COVID-19 infection a minimum of 3 months prior to contact with the study team
* Formal diagnosis of Long Covid from a physician
* Post-treatment Lyme disease syndrome
* Diagnosis will be based on participants meeting either Group 1 or Group 2 criteria of the Columbia Clinical Trial Network PTLDS diagnostic criteria:

  * Group 1. Well-defined Lyme disease meeting CDC Surveillance Definition Erythema Migrans History of possible exposure to a high incidence county or state (or an adjacent area) Erythema migrans rash

    * EM 1: EM rash diagnosed by HCP previously (either in person or telemedicine)
    * EM 1A: MOA self-report & medical record documentation of rash > 5 cm
    * EM 1B: MOA: self-report and medical record documentation of EM rash but not size
    * EM 1C: MOA: self-report & rash misdiagnosed in medical record as cellulitis/spider bite
    * EM 1D: MOA: self-report and either: photo of EM or Class 1 lab test confirmation within 4 weeks of illness onset OR
    * Disseminated "objective" manifestation with lab test confirmation of Bb infection
    * Clinical history includes at least one of the following symptoms/signs, which are not better accounted for by another cause (MOA: medical records and/or self-report).
    * Neurologic: Lymphocytic Meningitis ; Encephalitis; Encephalomyelitis Cranial Neuritis (especially facial palsy); Radiculoneuropathy; Other Neurologic Signs (with objective measures) : Encephalopathy, Polyneuropathy
    * Carditis: 2nd or 3rd degree AV block; Myocarditis; Pericarditis
    * Lyme arthritis: Recurrent joint swelling in one or more joints
    * Dermatologic: Disseminated EM ("satellite") or Acrodermatitis atrophicans AND
    * Lab test Confirmation (requires at least one of the Class 1 lab tests) (MOA: self-report & documentation)
  * Group 2. Probable

    * 2A. Chronic Multisystem Symptoms attributed to Lyme disease (insufficient to meet Group 1) and not better explained by another diagnosis and patient has evidence of positive lab results on a Class 1 lab test (or 4 of 10 bands for IgG Western blot (WB)) (MOA: self-report with lab documentation Class 1 lab test confirmation (excluding IgM WB) Highly suggestive IgG WB (4 of 10 bands) OR
    * 2B. EM rash by history after exposure to a Lyme-endemic area but not previously diagnosed by a HCP and no photo or Class 1 lab test confirmation is available (MOA: self-report) OR
    * 2C. Viral like illness (not better explained by other cause) with indeterminate or + enzyme immunoassay (EIA) with positive IgM WB or positive Class 1 lab test (within 4 weeks of illness onset after known exposure to a Lyme high-incidence area for standard two-tiered (STT) IgM) (MOA: medical records, lab test and self-report) (MOA: lab test and self-report) OR
    * 2D. Viral like illness (not better explained by other cause) with indeterminate or positive EIA with positive IgM WB or positive Class 1 lab test (within 6 months of illness onset after known exposure to a Lyme high-incidence area for standard two-tiered (STT) IgM)
* (MOA: medical records, lab test and self-report)
* (MOA: lab test and self-report)
* ME/CFS
* Formal diagnosis of ME/CFS prior to 2020 from a physician
* Actively symptomatic such that the 2011 International Criteria for ME/CFS is met at time of screening

Exclusion Criteria:

* Current use of antiplatelet or anticoagulation regimen
* Diagnosis of an autoimmune condition such as Chronic EBV, Multiple Sclerosis, Hashimoto's Disease, etc. which would impact the immunological profiling analysis.
* Pregnancy or lactation
* Known allergy to earthworms (Lumbrokinase is a supplement that is derived from earthworms)
* Past medical history of a bleeding or clotting disorder
* Has a scheduled surgery during, or immediately after, the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
EuroQol Visual Analogue Scale Score (EQ-VAS) | Up to 12 weeks
  The EQ VAS is a visual analogue scale that allows individuals to rate their overall health from 0 (worst imaginable health) to 100 (best imaginable health), providing a quantitative measure of health as judged by the patient.

SECONDARY OUTCOMES:
The EuroQol Five-Dimensional Health Questionnaire (EQ-5D-5L) | Up to 12 weeks
  The EQ-5D-5L is a validated, standardized, generic instrument that is a preference-based health- related quality of life questionnaire. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate their health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. Full scale from 5 to 25, with higher score indicating poorer health outcomes.
10-Meter Walk Test | Up to 12 weeks
  The scoring for the 10-meter walk test involves recording the time it takes to walk 10 meters and then calculating walking speed in meters per second (m/s). The test typically measures the time it takes to walk the middle 6 meters of a 10-meter walk, allowing for acceleration and deceleration.
Root mean square of successive differences between normal heartbeats (RMSSD) | Up to 12 weeks
  The RMSSD is obtained by first calculating each successive time difference between heartbeats in ms. Then, each of the values is squared and the result is averaged before the square root of the total is obtained. This is a measure of parasympathetic nervous system function. Higher RMSSD values generally indicate greater parasympathetic activity and a more resilient heart.
BrainCheck Cognitive Assessment Battery | Up to 12 weeks
  The BrainCheck software is an advanced digital cognitive assessment completed on a computer or tablet. Scores within one standard deviation of the mean are considered normal, while scores outside this range may suggest cognitive impairment.
General Symptom Questionnaire (GSQ-30) | Up to 12 weeks
  The General Symptom Questionnaire-30 (GSQ-30) is a valid and reliable instrument to assess symptom burden among patients with acute and post-treatment. The GSQ-30 total score ranges from 0 to 120, with higher scores indicating a greater symptom burden.
Medical Research Council Breathlessness Scale (MRC) | Up to 12 weeks
  The General Symptom Questionnaire-30 (GSQ-30) is a valid and reliable instrument to assess symptom burden among patients with acute and post-treatment. The GSQ-30 total score ranges from 0 to 120, with higher scores indicating a greater symptom burden.
Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) | Up to 12 weeks
  The Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) is a tool used to identify and classify pain, particularly neuropathic pain, based on a patient's reported symptoms and signs of nerve damage. A score of 12 or more on the LANSS is generally considered indicative of neuropathic pain.
Patient Health Questionnaire (PHQ-2) | Up to 12 weeks
  A PHQ-2 score ranges from 0 to 6, with 3 being the optimal cut-off point for depression screening. A score of 3 or higher indicates a high probability of major depressive disorder. A score of 2 or higher may be preferred in situations where clinicians want to ensure that few cases of depression are missed.
Generalized Anxiety Disorder (GAD-7) | Up to 12 weeks
  The GAD-7 is a 7-item scale developed and validated to identify generalized anxiety disorder and its severity. It assesses the frequency of 7 anxiety symptoms and scores the responses from 0 ("Not at all") to 3 ("Nearly every day"). Total scores of 5, 10, and 15 correspond to mild, moderate, and severe generalized anxiety disorder, respectively. Full scale from 0-21, with higher score indicating more symptoms.
Neuro-QoL™ v2.0 Cognitive Function-Short Form | Up to 12 weeks
  The Neuro-QoL Cognitive Function v2.0 short form assesses perceived difficulties in cognitive abilities, including memory, attention, decision making, planning, organizing, calculating, remembering, and learning. The short form consists of 8 questions assessed on a 5-point Likert scale, resulting in a raw score range of 8 to 40. A raw score is then converted to a T-score using conversion tables. Scores 0.5 - 1.0 SD worse than the mean (T-score 40-45) = mild symptoms/impairment. Scores 1.0 - 2.0 SD worse than the mean (T-score 30-40) = moderate symptoms/impairment. Scores 2.0 SD or more worse than the mean (T-score below 30) = severe symptoms/impairment.
Fatigue Severity Scale | Up to 12 weeks
  The Fatigue Severity Scale (FSS) uses a 7-point scale (1-7) to assess fatigue, with higher scores indicating greater severity, and a total score ranging from 9 to 63. Higher scores indicate more severe fatigue.
DePaul Post-Exertional Malaise Questionnaire (DSQ) | Up to 12 weeks
  The DSQ is designed to evaluate 54 classic ME/CFS symptoms, including fatigue, post-exertional malaise, sleep, pain, neurological/cognitive impairments, and autonomic, neuroendocrine, and immune symptoms. Each symptom's frequency and intensity are rated on a 5-point scale (0-4). Frequency and severity scores are multiplied by 25, added together, and then divided by 2 to create a composite frequency/severity score for each symptom. These scores range from 0 to 100, with higher scores indicating a greater symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: David Putrino, PhD, PT, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- The Cohen Center for Recovery from Complex Chronic Illnesses (CoRE), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No